CLINICAL TRIAL: NCT06064851
Title: Delivering Transcutaneous Auricular Neurostimulation to Reduce Heavy Menstrual Bleeding in Patients With and Without Von Willebrand Disease
Acronym: VWD/HMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Five Liters, Inc. (Industry)
Collaborators: Spark Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Organization: Spark Biomedical, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5L-BLD-05
Record Dates: First submitted 2023-09-15; First posted 2023-10-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Von Willebrand Disease, Type 1; Heavy Menstrual Bleeding
Keywords: Transcutaneous auricular vagus nerve stimulation; Neurostimulation; Hemostasis; Menstrual cycle; Menstruation; Blood loss; Hormone therapy; PBAC; Menorrhagia; CMSS
MeSH Terms: conditions — von Willebrand Disease, Type 1; Menorrhagia; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants with VWD and HMB will be enrolled in the study over the course of two consecutive menstrual cycles. First Menstruation will be baseline. Second Menstruation participants will self-administer 2, 1-hour sessions of active tAN daily beginning Day 1 of second menstruation through the final day of second menstruation.
Masking Description: No masking; open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Von Willebrand Disease (VWD) Patients (Experimental): Participants with VWD Type 1 who are on hormone therapy. First Menstruation (baseline/no active tAN) followed by Second Menstruation (active tAN)
  Interventions: Device: Volta System
- Heavy Menstrual Bleeding (HMB) Patients (Experimental): Participants with no known cause of HMB who are not on hormonal therapy. First Menstruation (baseline/no active tAN) followed by Second Menstruation (active tAN)
  Interventions: Device: Volta System

INTERVENTIONS:
Device: Volta System — The Volta System will be using the components of the Sparrow Ascent device: (FDA-cleared K230796) a wearable, battery-operated, neurostimulation system designed to transcutaneously stimulate nerves on and/or around the auricle. During Second Menstruation, participants will self-administer 2, 1-hour sessions of active tAN daily with the Volta System Device beginning Day 1 of second menstruation through the final day of second menstruation.

SUMMARY:
The objectives of this study are to determine if transcutaneous auricular neurostimulation (tAN) can modulate hemostasis, improve perceived quality of life, and improve pain during the menstrual cycle of von Willebrand Disease (VWD) patients.

DETAILED DESCRIPTION:
This study is designed as an open label, two-arm, decentralized clinical study in which patients with heavy menstrual bleeding (HMB) will receive tAN, which targets the auricular branch of the vagus nerve (ABVN) and the auriculotemporal nerve (ATN). Participants will be enrolled into one of two cohorts of the study over the course of two consecutive menstrual cycles.

1. Patients with VWD Type 1 who are on hormone therapy (n=15)
2. Patients with no known cause of HMB who are not currently on hormone therapy (n=15)

During the First Menstruation (baseline), no tAN treatment will be delivered. Participants will estimate blood loss daily throughout the duration of the menstruation phase of their first menstrual cycle. Dysmenorrhea, a general quality of life assessment, and total duration of menstruation will be collected on the final day of first menstruation.

During the Second Menstruation, participants will self-administer 2, 1-hour sessions (daily total of 2 hours) of active tAN daily beginning Day 1 of menstruation through the final day of second menstruation. Participants will estimate blood loss daily throughout the duration of the menstruation phase of their second menstruation. Dysmenorrhea, a general quality of life assessment, and total duration of menstruation will be collected on the final day of second menstruation.

ELIGIBILITY:
Inclusion Criteria:

1. Regularly menstruating female participants between 18-45 years of age
2. Typical length of menstruation ranging from 7 to 14 days
3. History of menorrhagia as assessed by the Menstrual Bleeding Questionnaire
4. For patients who have been diagnoses with von Willebrand Disease Type 1: On hormone therapy (with the exception of Nexplanon- at least three months) and willing to continue use for the duration of the study
5. For participants with idiopathic heavy menstrual bleeding: No use of hormon therapy for at least the past three months
6. No changes to all current medications and supplements in the past three months, willingness to continue use for duration of study, and not start any new medications or homeopathic remedies
7. Reliable access to an Internet-enabled device to complete required questionnaires
8. Willingness to consistently use the same brand of tampons and/or pads throughout duration of the study

Exclusion Criteria:

1. Pregnancy within three months of enrollment
2. Lactating at the time of enrollment
3. Antifibrinolytic use within 30 days of enrollment
4. Acquired bleeding disorder
5. Use of anticoagulants (i.e., Aspirin, Warfarin, Coumadin, etc.) including platelet inhibitors for 30 days prior to enrollment
6. Use of the Copper intrauterine device within the past 3 months
7. Known structural cause of heavy menstrual bleeding
8. Use of menstrual cups as a method of menstrual blood collection
9. Participant has a history of chronic tobacco use or has ingested nicotine via smoking, vaping, smokeless tobacco, or nicotine patches in the past three months
10. Participant has received a blood transfusion within 30 days prior to study
11. Participant has a history of epileptic seizures
12. Participant has a history of neurologic diseases or traumatic brain injury
13. Participant has presence of devices (e.g., pacemakers, cochlear prostheses, neurostimulators)
14. Participant has abnormal ear anatomy or ear infection present
15. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants are risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Regularly menstruating female participants.
Enrollment: 29 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Blood loss during menses in both groups | Daily throughout both menstruations (up to 2 complete menstrual cycles- estimated 60 days)
  Comparison of mean Pictorial Bleeding Assessment Chart (PBAC) scores during first menstruation (no stimulation) versus second menstruation (active stimulation). The PBAC is a widely accepted tool for patients with HMB to account for menstrual blood loss. Menstrual blood loss is estimated through a selection of images of tampons, pads, clots, and flooding events. Patients mark a tally next to the images that best match each of the menstruation products they used that day. This trial will utilize a modified version of the Wyatt et al. 2001 PBAC, where a tally system will be added to each of the images.
Quality of Life in both groups | Final day of each menstruation (up to 2 complete menstrual cycles- estimated 60 days)
  Comparison of mean quality of life score measured by the Short Form 36 (SF-36) during first menstruation (no stimulation) versus second menstruation (active stimulation). The SF-36 is a 36-item patient-reported questionnaire that assesses general quality of life. This questionnaire includes eight variables: physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy and vitality, pain, and general perception of health. The SF-36 is scored using a standardized scoring algorithm or by the SF-36 scoring software. The SF-36 scores range from 0 to 100, with higher scores representing better health status.
Duration and severity of dysmenorrhea in both groups | Final day of each menstruation (up to 2 complete menstrual cycles- estimated 60 days)
  Comparison of mean Cox Menstrual Symptom Scale (CMSS) scores during first menstruation (no stimulation) versus second menstruation (active stimulation). The CMSS measures menstrual distress and dysmenorrhea. The CMSS Severity subscale is an 18-item self-reported scale that measures severity of menstrual symptoms, including pain, nausea, emotions, etc. during menstruation. The CMSS will be used in this trial to measure a participant's dysmenorrhea every day of each menstruation. Each CMSS item is scored from 0-4, with a higher score indicating higher dysmenorrhea severity.
Duration of menstruation in both groups | Final day of each menstruation (up to 2 complete menstrual cycles- estimated 60 days)
  Compare duration of menstruation between first menstruation (no stimulation) versus second menstruation (active stimulation).

CONTACTS AND LOCATIONS:
Overall Officials: Navid Khodaparast, PhD, Principal Investigator — Chief Science Officer; Melanie McWade, PhD, Study Director — Senior Director of Clinical Operations
Locations (1):
- Five Liters, Dallas, Texas, United States